CLINICAL TRIAL: NCT05777824
Title: Pathological Response Adapted Decision-making of Postoperative Management for HNSCC Receiving Induction Immunotherapy and Chemotherapy
Brief Title: Postoperative Management for HNSCC Based on Pathological Response of Induction Chemotherapy and Immunotherapy
Acronym: HN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22/523-3725
Record Dates: First submitted 2023-03-07; First posted 2023-03-21 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-02

CONDITIONS: Head and Neck Cancer
Keywords: postoperative radiotherapy; induction immunotherapy and chemotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- low-risk and PCR (No Intervention): Observation
- low-risk and MPR (Experimental): immunotherapy maintenance
  Interventions: Combination Product: anti-PD-1 or PD-L1 antibody
- low-risk and IPR (Experimental): postoperative radiotherapy (50 Gy) and immunotherapy maintenance
  Interventions: Combination Product: anti-PD-1 or PD-L1 antibody; Radiation: postoperative radiaotherapy
- high-risk and PCR (Experimental): postoperative radiotherapy (50 Gy) and immunotherapy maintenance
  Interventions: Combination Product: anti-PD-1 or PD-L1 antibody; Radiation: postoperative radiaotherapy
- high-risk and MPR (Experimental): postoperative radiotherapy (60 Gy) and immunotherapy maintenance
  Interventions: Combination Product: anti-PD-1 or PD-L1 antibody; Radiation: postoperative radiaotherapy
- high-risk and IPR (Experimental): postoperative concurrent chemoradiotherapy (60 Gy) and immunotherapy maintenance
  Interventions: Combination Product: anti-PD-1 or PD-L1 antibody; Radiation: postoperative radiaotherapy

INTERVENTIONS:
Combination Product: anti-PD-1 or PD-L1 antibody — immunotherapy maintenance with anti-PD-1 or PD-L1 antibody every three weeks for 13 cycles after radiotherapy
  Arms: high-risk and IPR; high-risk and MPR; high-risk and PCR; low-risk and IPR; low-risk and MPR
Radiation: postoperative radiaotherapy — postoperative radiotherapy (60Gy or 50Gy)
  Arms: high-risk and IPR; high-risk and MPR; high-risk and PCR; low-risk and IPR

SUMMARY:
To develop postoperative stratification treatment for patients who have received induction chemotherapy and immunotherapy in locally advanced head and neck cancers. Risk stratification is based on clinical characteristics and pathological responses. In order to achieve no inferior survival rate and a lower treatment-related toxicity rate than the standard treatment.

DETAILED DESCRIPTION:
Induction chemotherapy combined with immunotherapy has shown promising efficacy in the treatment of patients with locally advanced head and neck cancers. However, how to choose a proper postoperative treatment remains unknown. Eligibility patients were assigned to two arms, each divided into three groups: observation, immunotherapy maintenance, and radiotherapy (50 Gy dose) plus immunotherapy maintenance group for low-risk arm; radiotherapy (50 Gy or 60Gy dose) plus immunotherapy maintenance groups, concurrent chemotherapy plus immunotherapy maintenance group for a high-risk arm. Disease-free survival, overall survival, and treatment-related toxicity would be calculated to evaluate the efficacy of treatments.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects are not limited by gender, age from 18 to 75 years old;
2. Histopathologically confirmed squamous cell carcinoma of the head and neck cancer;
3. Locally advanced squamous cell carcinoma diagnosed as T3-4 or N+ stage according to AJCC 8th edition staging;
4. ECOG score 0-1;
5. without distant metastasis;
6. received induction chemotherapy plus immunotherapy, followed by surgery
7. The expected survival is expected to be no less than 6 months.
8. No contraindications to chemotherapy, immunotherapy, and radiotherapy;

Exclusion Criteria:

1. Past malignancies history (except for stage I non-melanoma skin cancer or cervical carcinoma in situ)
2. Received any systemic anti-tumor therapy for target lesions before induction chemotherapy and immunotherapy;
3. Previously experienced head and neck radiation therapy;
4. Subjects who have used corticosteroids (>10 mg/day prednisone or other equivalent hormones) or other immunosuppressive agents for systemic treatment within 1 month before enrollment. In the absence of active autoimmune disease, inhaled or topical corticosteroids and adrenal hormone replacement therapy at therapeutic doses of prednisone ≤10 mg/day are permitted;
5. Patients with pleural effusion, pericardial effusion or ascites that need to be drained with clinical symptoms, or who have received serous cavity effusion drainage for the purpose of treatment within 2 weeks before enrollment;
6. Severe comorbidities including myocardial infarction, arrhythmia, cerebral vascular disease, ulceration disease, mental disease and uncontrolled diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 2 years
  defined as the time from random assignment to documented local or regional relapse, distant metastasis, or death from any cause, whichever occurred first after 2 years of treatment.

SECONDARY OUTCOMES:
Overall survival | 2 years
  defined as the time from random assignment to death from any cause or censored at the date of last follow-up.
Local-Regional failure survival | 2 years
  defined as the time from random assignment to documented local or regional relapse, whichever occurred first after 2 years of treatment.
Toxicity Adverse events | 2 years
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events (acute toxicity) and late radiation toxicities were assessed by NCI-CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Junlin Yi, Doctor, Study Chair — National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, CAMS & PUMC
Locations (1):
- National Cancer Center /National Clinical Research Center for Cancer/Cancer Hospital, CAMS & PUMC, Beijin, Beijing Municipality, China